CLINICAL TRIAL: NCT06764563
Title: The Effect of a Mediterranean Diet on Quality of Life in Multiple Sclerosis Patients
Acronym: Mediet4MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Ariel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TLV-0621-23
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; mediterranean diet; quality of life
MeSH Terms: conditions — Multiple Sclerosis | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: Block randomize assignment to two study groups: intervention and control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention- Mediterranean diet nutritional counselling (Experimental)
  Interventions: Behavioral: Mediterranean Medical Nutrition Therapy (counselling)
- control, no dietary change (No Intervention): Participants in the non-dietary intervention group will continue their usual diet

INTERVENTIONS:
Behavioral: Mediterranean Medical Nutrition Therapy (counselling) — The participants in the intervention group will receive dietary guidance on the Mediterranean diet during 9 sessions over six months. The sessions which will be held in groups of ten individuals. In-person group sessions will be held three times: at the first meeting, after three months, and after six months. During the remaining six sessions, 6 online video sessions (by the institutional telemedicine program) will be delivered and include 60 minutes of nutritional educational sessions with a registered dietitian once a month
  Arms: Intervention- Mediterranean diet nutritional counselling

SUMMARY:
The role of dietary interventions in improving symptoms of multiple sclerosis (MS) is of high interest amongst patients and researchers, but data supporting this evidence are limited. Current evidence indicates that A higher Expanded Disability Status Scale (EDSS) score correlates with poor diet quality in patients with MS. Moreover, even though disease-modifying therapies (DMT) improve disease course and prognosis, MS patients report a lower quality of life (QoL) than people without illness. The Mediterranean diet (Med-Diet) is beneficial in preventing cardiovascular comorbidities, and outcomes of a decrease in inflammation processes are evident. Recent studies suggest that the Med-Diet might positively affect MS QoL, However, empirical evidence remains unclear, limiting the possibility of evidence-based nutritional recommendations. In the current study, we aim to investigate the effect of the Mediterranean diet on the quality of life of patients with MS.

Methods:

Randomized controlled trial among MS patients aged 18-70. The participants will be randomly assigned to two 1:1 ratio groups: The med-diet group and the control group (no intervention). The intervention will be carried out for six months with subsequent six-months follow-up.

Nine nutrition sessions will be delivered to the intervention group by an expert registered clinical dietitian. Data will be collected at baseline, three months, six months, and 12 months, including the following: Demographic, Anthropometric measurements, Blood tests of complete blood count, chemistry, levels of vitamins D, and B12, CRP, neurofilaments light chain (NfL), Grip strength, Biochemical analysis for fatty acid composition in membranes of red blood cells (RBC) and HPLC analysis of carotenoid concentration. Patients will complete questionnaires for multiple sclerosis quality of life-54 (MSQoL-54), Patient Health Questionnaire (PHQ-9), Fatigue Severity Scale Questionnaire (FSS) and will undergo clinical evaluation for expanded disability status scales (EDSS) and Symbol Digit Modalities Test (SDMT). Dietary analysis and Med-Diet adherence will be validated by the Israeli Mediterranean diet screener (I-MEDAS) and by Food diaries.

Calculated sample size: To achieve a mean difference of 10 points in the MSQoL-54 questionnaire and 80% power, a sample of 77 participants per group is needed. Considering a 5% drop-off, 81 participants per group are needed, and overall, 162 participants.

Expected results: this study will highlight the effect of the Med-Diet dietary pattern on MS quality of life, MS symptoms, and its underlying mechanism, to enable evidence-based nutritional recommendations for MS patients

Importance to Medicine: MS patients suffer from a decrease in QoL. Hence, physicians, researchers, and patients seek nutritional approaches that may improve their condition. If proven beneficial, The Med diet, a dietary approach that has been proven to reduce the risk for major comorbidities and that can be sustained throughout life, has the potential to improve the condition of MS patients in crucial lifestyle aspects.

DETAILED DESCRIPTION:
Currently, there is no definite cure for MS. The current treatments may slow down the degree of disease activity and improve the prognosis of the patients. Yet, still many patients suffer from a decrease in the QoL. The lack of a cure and the reduced QOL raise interest among patients, physicians, and researchers regarding nutritional approaches that may improve the condition of the patients . Indeed, a higher EDSS score has been correlated with poor diet quality. The Western diet, characterized by a high intake of saturated fats, omega-6 fatty acids, and a high proportion of refined carbohydrates, may lead to the activation of pro-inflammatory immune pathways and is therefore not recommended. The Med-Diet is beneficial in preventing heart diseases, and outcomes of a decrease in inflammation processes are evident .Thus, the Med-Diet might have an additive beneficial effect with the current disease-modifying drugs (DMTs) in improving disease severity . Furthermore, the Med-Diet is easy for lifelong adherence compared to the various diets investigated in MS (e.g., ketogenic diets, gluten-free, very low-fat, and fasting-mimicking diets), which require careful clinical monitoring . In addition, Recent studies have shown that the Med-Diet positively affects MS fatigue . Whereas people with MS (pwMS) are highly interested in diet as a potential protective factor against disability and improving QOL and other MS symptoms , empirical evidence remains unclear, limiting the possibility of evidence-based nutritional recommendations. Finally, even though the Med-Diet is known for its anti-inflammatory effect, its exact mechanism and effect on MS progression are still not fully understood. Hence, this study will highlight the potential effects and pathways of Med-Diet to improve the QoL of MS patients.

1. Study Design: A single-blind, randomized controlled, single-center study.

   1. MS patients, men and women, Aged 18-70 with confirmed MS diagnosis based on 2017 Mcdonald criteria, fulfilling the eligibility criteria.
   2. Baseline data (Time 0 - T0) Socioeconomic and lifestyle information on smoking, physical activity, and medical information regarding disease type and activity. Moreover, Baseline, three months, six months, and 12-month (T0, T3, T6, T12) assessments of: questionnaires: Mediterranean adherence diet questionnaire (I- MEDAS), MS Quality of Life-54 (MSQoL-54), Patient Health Questionnaire (PHQ-9), Fatigue Severity Scale Questionnaire (FSS). Anthropometric measurements: height, weight, waist circumference, bioelectrical impedance analysis, including fat mass and fat-free mass, Hand grip strength. Clinical assessment: A note on the appearance of relapses from the previous visit, EDSS, SDMT, Blood test for complete blood count, chemistry, levels of vitamins D and vitamin B12, CRP, fatty acid composition in red blood cell membranes , neurofilament light chain (NfL), and carotenoids plasma concentration. Food intake will be measured using food diaries, adherence to Med-Diet will be measured using the I-MEDAS .
   3. Length of intervention- 6 months. Follow-up will occur immediately after the intervention (T6) and 6 months after the intervention (T12). The main outcome variable will be QOL as measured by the MSQoL-54 questionnaire.
   4. The interventions will occur in the Neuroimmunology and Multiple Sclerosis Unit at Tel Aviv Sourasky Medical Center.
2. Methods (Sample size and its justification should be included & available equipment/means)

   1. All eligible patients fulfilling the eligibility criteria will be contacted by study personnel after approval from the treating physician and asked to come for a baseline meeting and explanation of study procedures. Those meeting all inclusion criteria and willing to provide informed consent will be enrolled.
   2. Randomization: Individuals will be randomized to intervention or control groups by stratified randomization, where the stratification will be by the severity of the disease as measured by EDSS ( EDSS ≤3, EDSS>3) and sex. To obtain population representativeness and based on the difference between sexes in the disease prevalence, participants will be randomized separately with a ratio of two women per man in the study.
   3. Sample size: Based on the average score (mean±SD) of 58.2±21.9 detected in the QoL54 MS questionnaire, to achieve a mean difference between the groups of 10 points in the questionnaire and 80% power, a sample of 77 participants per group is needed. With an anticipated discontinuation/dropout rate, 81 participants per group are needed overall 162 participants
   4. Statistical analysis: The investigators will further be able to ensure sufficient power for a multivariate regression model according to the following criteria: The model will include four covariates, which will yield an R-squared of at least .070. It will include one variable (study group), which will yield an increment of .050. The total R-squared for the five variables in the model will be at least .120. With the given sample size of 160 and alpha set at .05, the study will have a power of 0.84

ELIGIBILITY:
Inclusion Criteria:

* Confirmed MS based on 2017 Mcdonald criteria, with stable medication regimen in the previous six months.

Exclusion Criteria:

* Pregnancy or lactating
* People with a lack of judgment
* Serum creatinine ≥2 mg/dL(177 μmol per liter) or more
* Patients who had gastrointestinal problems that would prevent them from following any of the test diets
* Patients who had liver dysfunction (an increase by a factor of at least two above the upper limit of normal in alanine aminotransferase and aspartate aminotransferase levels)
* Active cancer or chemotherapy treatment in the last three years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
MS QOL score | six months
  As measured in MSQOL-54 questionnaire. score range 0-100. Higher score mean a better outcome.

SECONDARY OUTCOMES:
Disease Disability score | six months
  Decrease in Expanded disability status scale (EDSS) score. Range between 0-10. Higher score mean worse outcome
Chronic fatigue levels | Six months
  Fatigue Severity Scale (FSS) questionnaire score. Range of score between 1-7. Higher score mean worse outcome.
Depression levels | six months
  As measured in PHQ-9 Questionnaire. Score range between: 0-27. Higher score mean worse outcome.
Carotenoid plasma concentration. | six months
Neurofilament light chain (NfL). | six months
  As measured in blood plasma
Cognitive function | six months
  increase in Symbol Digit Modalities Test (SDMT).

OTHER OUTCOMES:
Vitamin B12 | six months
  As measured in blood plasma
Body Mass Index (BMI) | six months
  Measured in kg/m2
Muscle strength | six months
  As measured by JAMAR hand grip
Low density lipoprotein levels (LDL) | six months
  As measures in blood plasma
CRP levels | six months
  As measured in blood serum
Vitamin D levels | six months
  As measured in blood plasma
Height | six months
  As measured in meters
Weight | six months
  Measured in kg
Waist circumference | six months
  As measured in cm
High density lipoprotein levels (HDL) | six months
  As measured in blood plasma
Triglycerides | six months
  As measured in blood plasma
Muscle Mass | six months
  As measured with Bioimpedance scale in kg
Fat mass | six months
  As measured in bioimpedance scale in percentages
Fatty acid composition in red blood cells membrane | Six months
  As measured

CONTACTS AND LOCATIONS:
Overall Officials: Vered Kaufman-Shriqui, PhD, Principal Investigator — Ariel University
Locations (1):
- Tel Aviv Sourasky medical center, Tel Aviv, Israel, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghasemi N, Razavi S, Nikzad E. Multiple Sclerosis: Pathogenesis, Symptoms, Diagnoses and Cell-Based Therapy. Cell J. 2017 Apr-Jun;19(1):1-10. doi: 10.22074/cellj.2016.4867. Epub 2016 Dec 21. PMID 28367411
- [Background] Swank RL, Dugan BB. Effect of low saturated fat diet in early and late cases of multiple sclerosis. Lancet. 1990 Jul 7;336(8706):37-9. doi: 10.1016/0140-6736(90)91533-g. PMID 1973220
- [Background] Yu M, Jelinek G, Simpson-Yap S, Neate S, Nag N. Self-reported ongoing adherence to diet is associated with lower depression, fatigue, and disability, in people with multiple sclerosis. Front Nutr. 2023 Mar 1;10:979380. doi: 10.3389/fnut.2023.979380. eCollection 2023. PMID 36937366
- [Background] Shai I, Spence JD, Schwarzfuchs D, Henkin Y, Parraga G, Rudich A, Fenster A, Mallett C, Liel-Cohen N, Tirosh A, Bolotin A, Thiery J, Fiedler GM, Bluher M, Stumvoll M, Stampfer MJ; DIRECT Group. Dietary intervention to reverse carotid atherosclerosis. Circulation. 2010 Mar 16;121(10):1200-8. doi: 10.1161/CIRCULATIONAHA.109.879254. Epub 2010 Mar 1. PMID 20194883
- [Background] Mousavi-Shirazi-Fard Z, Mazloom Z, Izadi S, Fararouei M. The effects of modified anti-inflammatory diet on fatigue, quality of life, and inflammatory biomarkers in relapsing-remitting multiple sclerosis patients: a randomized clinical trial. Int J Neurosci. 2021 Jul;131(7):657-665. doi: 10.1080/00207454.2020.1750398. Epub 2020 Apr 16. PMID 32249637
- [Background] Moravejolahkami AR, Paknahad Z, Chitsaz A. Association of dietary patterns with systemic inflammation, quality of life, disease severity, relapse rate, severity of fatigue and anthropometric measurements in MS patients. Nutr Neurosci. 2020 Dec;23(12):920-930. doi: 10.1080/1028415X.2019.1580831. Epub 2019 Mar 21. PMID 30896320
- [Background] Evans E, Levasseur V, Cross AH, Piccio L. An overview of the current state of evidence for the role of specific diets in multiple sclerosis. Mult Scler Relat Disord. 2019 Nov;36:101393. doi: 10.1016/j.msard.2019.101393. Epub 2019 Sep 9. PMID 31574403
- [Background] Katz Sand I, Benn EKT, Fabian M, Fitzgerald KC, Digga E, Deshpande R, Miller A, Gallo S, Arab L. Randomized-controlled trial of a modified Mediterranean dietary program for multiple sclerosis: A pilot study. Mult Scler Relat Disord. 2019 Nov;36:101403. doi: 10.1016/j.msard.2019.101403. Epub 2019 Sep 24. PMID 31610401